CLINICAL TRIAL: NCT06836505
Title: Safety and Efficacy of CAR-T Cell Therapy for Relapsed/refractory Neuroblastoma and Desmoplastic Small Round Cell Tumors: a Single-arm, Open-label Trial.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry); Dongguan Taixin Hospital (Unknown)
Responsible Party: Principal Investigator, Yizhuo Zhang, professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXEC-2024-025
Record Dates: First submitted 2025-01-25; First posted 2025-02-20 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-12

CONDITIONS: Neuroblastoma (NB); Desmoplastic Small Round Cell Tumor (DSRCT)
Keywords: CART, Neuroblastoma, Desmoplastic Small Round Cell Tumor
MeSH Terms: conditions — Neuroblastoma; Desmoplastic Small Round Cell Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Safety and efficacy of CAR-T cell therapy for relapsed/refractory NB and DSRCT (Experimental)
  Interventions: Biological: CART therapy

INTERVENTIONS:
Biological: CART therapy — GD2/B7H3 CAR T-cell therapy

SUMMARY:
Title: Safety and efficacy of CAR-T cell therapy for relapsed/refractory neuroblastoma and desmoplastic small round cell tumors: a single-arm, open-label trial.

The CART used in this study will be provided by Shanghai YaKe Biotechnology Ltd.

Aims:

1. To evaluate the safety and efficacy of GD2/B7H3 CAR-T therapy for relapsed/refractory neuroblastoma, and observe its pharmacokinetic/pharmacodynamic characteristics and the survival of CAR-T cells in relapsed/refractory neuroblastoma patients.
2. To evaluate the safety and efficacy of GD2/B7H3 CAR-T therapy for relapsed/refractory desmoplastic small round cell tumor, and observe its pharmacokinetic/pharmacodynamic characteristics and the survival of CAR-T cells in desmoplastic small round cell tumor patients.

Patients: Relapsed/refractory neuroblastoma; Relapsed/refractory desmoplastic small round cell tumor.

CAR-T therapy: Lymphodepletion treatment will be performed within 14 days prior to CAR-T cell infusion: intravenous chemotherapy based on fludarabine 25mg/m² and cyclophosphamide 500mg/m² for 1 to 3 days. CAR-T cells will then be infused intravenously, with a dosage of 1.00 to 10.00 × 10⁶/kg of CAR-positive T cells.

Research period: CAR-T cell infusion will be followed up for one year, or until adverse events resolve, progression occurs, or the patient transitions to other treatments.

Outcome measures:

Incidence of adverse events related to CAR-T therapy, as well as their intensity and duration; Pharmacokinetic/pharmacodynamic characteristics of CAR-T in patients and the survival of CAR-T cells.

Overall response rate (ORR) after CAR-T cell infusion, including complete response (CR) and partial response (PR); Overall survival (OS), progression-free survival (PFS), event-free survival (EFS), time to progression (TTP), and duration of response (DOR) after CAR-T cell infusion;

DETAILED DESCRIPTION:
Main objective:

To evaluate the safety, pharmacokinetic/pharmacodynamic characteristics and the survival of CAR-T cells in relapsed/refractory neuroblastoma and desmoplastic small round cell tumor patients.

Secondary objectives:

To evaluate the efficacy of CAR-T cells in relapsed/refractory neuroblastoma and desmoplastic small round cell tumor patients.

Patients: Relapsed/refractory neuroblastoma; Relapsed/refractory desmoplastic small round cell tumor.

CAR-T therapy: Lymphodepletion treatment will be performed within 14 days prior to CAR-T cell infusion: intravenous chemotherapy based on fludarabine 25mg/m² and cyclophosphamide 500mg/m² for 1 to 3 days. CAR-T cells will then be infused intravenously, with a dosage of 1.00 to 10.00 × 10⁶/kg of CAR-positive T cells.

Research period: CAR-T cell infusion will be followed up for one year, or until adverse events resolve, progression occurs, or the patient transitions to other treatments.

Outcome measures:

Incidence of adverse events related to CAR-T therapy, as well as their intensity and duration; Pharmacokinetic/pharmacodynamic characteristics of CAR-T in patients and the survival of CAR-T cells.

Overall response rate (ORR) after CAR-T cell infusion, including complete response (CR) and partial response (PR); Overall survival (OS), progression-free survival (PFS), event-free survival (EFS), time to progression (TTP), and duration of response (DOR) after CAR-T cell infusion;

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed as relapsed/refractory neuroblastoma or relapsed/refractory desmoplastic small round cell tumors;
2. Age 1-50 years, any gender;
3. Agree to participate in the trial and sign a written informed consent form;
4. Expected survival of ≥12 weeks;
5. Karnofsky performance status (for patients ≥16 years) or Lansky performance status (for patients <16 years) (Appendix 1) must be at least 50;
6. Good function of major organs:

   1. Liver function: ALT ≤ 5 times the upper limit of normal for the corresponding age, and bilirubin ≤ 2.0 mg/dL, except for patients with Gilbert-Meulengracht syndrome. Patients with Gilbert-Meulengracht syndrome who have bilirubin ≤ 3.0 times the upper limit of normal and direct bilirubin ≤ 1.5 times the upper limit of normal may be included;
   2. Renal function: Plasma creatinine ≤ 1.5 times the upper limit of normal, or estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73m²;
   3. Pulmonary function: Oxygen saturation ≥ 95% in room air;
   4. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 45%;
7. Patients using the following medications must meet the following conditions:

   Steroids: Steroid treatment doses must be stopped at least 2 weeks before CAR-T infusion. However, physiological replacement doses of steroids are allowed; Immunosuppressants: Any immunosuppressive drugs must be stopped at least 4 weeks before enrollment; Anti-proliferative treatments other than lymphodepleting chemotherapy within two weeks before infusion; CNS disease prophylaxis must be stopped 1 week prior to CAR-T infusion (e.g., intrathecal methotrexate injection);
8. Patients of childbearing potential (both male and female) must agree to use reliable contraception methods (hormonal or barrier methods or abstinence) with their partner until at least 12 months after CAR-T cell infusion, and until two consecutive flow cytometry or PCR tests show no CAR-T cells in the body;
9. If the subject cannot provide suitable T cells for CAR-T preparation, T cells from a healthy donor may be collected for preparation.

Exclusion Criteria:

* Patients with any of the following items will not be enrolled in this study:

  1. Patients with increased intracranial pressure or altered consciousness;
  2. Patients who have received radiation therapy within 2 weeks prior to infusion;
  3. Patients with active hepatitis B (defined as HBV DNA > 500 IU/mL) or hepatitis C (HCV RNA positive);
  4. HIV-positive patients or patients with a positive syphilis test;
  5. Patients with uncontrolled acute life-threatening bacterial, viral, or fungal infections (e.g., positive blood cultures within ≤72 hours before infusion);
  6. Patients with unstable angina and/or myocardial infarction within 6 months prior to screening;
  7. Patients with a history of or concurrent malignancies, except for the following conditions:

     1. Basal cell carcinoma or squamous cell carcinoma that has been adequately treated (sufficient wound healing required before study enrollment);
     2. Carcinoma in situ of the cervix or breast that has been cured, with no signs of recurrence for at least 3 years before the study;
     3. Primary malignant tumors that have been completely resected and have been in complete remission for ≥5 years;
  8. Pregnant or breastfeeding female patients;
  9. Patients with uncontrolled arrhythmias that have not been managed medically;
  10. Patients who need oral anticoagulation therapy within 1 week before CAR-T cell infusion;
  11. Patients with active neuroautoimmune or inflammatory diseases (e.g., Guillain-Barré syndrome, amyotrophic lateral sclerosis);
  12. Other conditions deemed inappropriate for participation in the clinical study by the investigator.

Patients enrolled in the clinical study must meet the inclusion criteria and not meet the exclusion criteria.

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-12-12 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of CAR-T cells in relapsed/refractory neuroblastoma and desmoplastic small round cell tumor patients. | From enrollment to the end of treatment at 1 year
  1. To evaluate the safety of the infusion of CAR T cells at different escalating/deescalating doses and establish the dose limiting toxicity (DLT) of the cellular product. Toxicity will be evaluated according to the CTC AE scale, version 4.0. DLT will be defined as any of the following that is not pre-existing, due to infection or to underlying malignancy and that may be considered possibly, probably or definitely related to the study cellular products. (1) Non-hematologic DLT is any grade 3 or 4 non-hematologic toxicity; (2) Hematologic DLT is defined as any grade 4 hematologic toxicity related to infusion ; (3) Grade 4 reactions related to infusion; (4) Death related to CAR T cells infusions.
     The incidence of grade 3-5 toxicities, with a main attention to severe Cytokine Release Syndrome (CRS), will be evaluated.
  2. To determine the optimal dose of CAR transduced T cells resulting in the control of the disease without inducing unacceptable levels of toxicity (MTD) .

SECONDARY OUTCOMES:
To evaluate the efficacy of CAR-T cells in relapsed/refractory neuroblastoma and desmoplastic small round cell tumor patients. | From enrollment to the end of treatment at 1 year
  To assess the antitumor effect of iC9-GD2-CAR T cells at 6 weeks, 3 and 6 months post-infusion. The Best Overall Response Rate (BOR) and the proportion of neuroblastoma patients achieving complete remission (CR) will be assessed according to INRC. The Best Overall Response Rate (BOR) and the proportion of desmoplastic small round cell tumor patients achieving complete remission (CR) will be assessed according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Dongguan Taixin Hospital, Dongguan, Guang
  - Shanghai YaKe Biotechnology Ltd., Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No